CLINICAL TRIAL: NCT00713336
Title: A Phase I, Double-blind, Double-dummy, Placebo-controlled, Randomised, Four-period Crossover Study to Assess the Effects of Single Oral Doses of ZD4054 (Zibotentan) (10mg and 30mg) on QTc Interval Compared to Placebo, Using AVELOX (Moxifloxacin) as a Positive Control, in Healthy Volunteers Aged 18 to 45 Years.
Brief Title: Four-period Crossover Study to Assess the Effects of Single Oral Doses of ZD4054 (Zibotentan) (10mg and 30mg) on QTc Interval
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr Thomas Morris, Medical Science Director, AstraZeneca, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: D4320C00017; ZD4054IL0017
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: ZD4054; Healthy Volunteers; QT interval
MeSH Terms: interventions — ZD4054; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): ZD4054 + Moxifloxacin placebo
  Interventions: Drug: ZD4054; Drug: Moxifloxacin placebo
- 2 (Active Comparator): ZD4054 placebo + Moxifloxacin
  Interventions: Drug: ZD4054; Drug: Moxifloxacin; Drug: ZD4054 Placebo
- 3 (Experimental): ZD4054 + ZD4054 placebo + Moxifloxacin placebo
  Interventions: Drug: ZD4054; Drug: Moxifloxacin placebo; Drug: ZD4054 Placebo
- 4 (Placebo Comparator): ZD4054 Placebo + Moxifloxacin placebo
  Interventions: Drug: ZD4054; Drug: ZD4054 Placebo; Drug: Moxifloxacin placebo

INTERVENTIONS:
Drug: ZD4054 — ZD4054 10mg Tablet
  Other Names: Zibotentan
Drug: Moxifloxacin — 400 mg capsule
  Other Names: AVELOX
  Arms: 2
Drug: ZD4054 Placebo — 3 tablets
  Arms: 2; 4
Drug: Moxifloxacin placebo — 1 capsule
  Arms: 1; 3; 4
Drug: ZD4054 Placebo — 2 tablets
  Arms: 3
Drug: ZD4054 — 30mg tablet
  Arms: 1
Drug: ZD4054 — 10mg tablet
  Arms: 3

SUMMARY:
This Study compares two ZD4054 (Zibotentan) doses (10mg and 30mg) with a placebo and a positive control to look at ZD4054 (Zibotentan)'s effect on the ECG of Healthy Volunteer

ELIGIBILITY:
Inclusion Criteria:

* Non Smoker
* Normal resting 12-lead ECG with normal QTc interval (<450 msec)
* Negative screens for serum hepatitis B surface antigen, hepatitis C antibody and Human Immunodeficiency Virus (HIV) at screening

Exclusion Criteria:

* Receipt of another new chemical entity in the 4 months before dosing in this study; participation in another study and participation in a non-invasive methodology study in which no drugs were given within 30 days before dosing in this study
* Risk (in the investigator's opinion) of transmitting, through blood or other body fluids, the agents responsible for acquired immune deficiency syndrome (AIDS), hepatitis B or hepatitis C
* Judgement by the investigator, that the healthy volunteer should not participate in the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-06; Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
to assess the maximum of the mean changes in time-matched QTcX (study specific correction) intervals after ZD4054 (Zibotentan) administration (10mg and 30mg) compared to placebo | Pre-dose, 0.5hr, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h

SECONDARY OUTCOMES:
assess the maximum of the mean changes in time-matched QT, QTcB (Bazett's correction), QTcF (Fridericia's correction) and QTcI (subject specific correction) intervals after ZD4054 (Zibotentan) administration (10mg and 30mg) compared to placebo | Pre-dose, 0.5hr, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h
assess the maximum of mean changes in time-matched QTcX, QT, QTcB, QTcF and QTcI intervals after moxifloxacin administration compared to placebo. | Pre-dose, 0.5hr, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h
further assess the safety and tolerability of ZD4054 (Zibotentan) by assessment of adverse events (AEs), laboratory variables and vital signs. | From time of Consent to Last Follow-up Visit

CONTACTS AND LOCATIONS:
Overall Officials: Raj Chetty, MD, Principal Investigator — Clinical Pharmacology UnitAlderley ParkAstraZenecaMacclesfieldSK10 4TG
Locations (1):
- Research Site, Macclesfield, United Kingdom